CLINICAL TRIAL: NCT06351722
Title: Effect of Non-surgical Periodontal Treatment in Smokers on SIRT-1 and Proteins of the NLRP3 Inflammasome and Long Noncoding RNAs
Brief Title: Non-surgical Periodontal Treatment in Smokers on SIRT-1, NLRP3 Inflammasome and LncRNAs
Status: Not yet recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zeynep Tastan Eroglu, assistant professor, Necmettin Erbakan University
Other Study IDs: smokingnlrp3inflasome
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Periodontitis, Adult
Keywords: periodontitis; smoking; NLRP3 inflammasome; SIRT1; non-coding RNA
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Serum, white cells and saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Non-smoking periodontitis (NSP): participants who reported never smoking, with clinical attachment loss ≥3 mm in >30% of sites, with probing depth ≥5 mm in at least six teeth, and with radiographic bone loss extending to or beyond the middle third of the root in the coronal third will be included.
  Interventions: Diagnostic Test: Before non-surgical periodontal treatment; Procedure: non-surgical periodontal treatment; Diagnostic Test: 3rd month after non-surgical periodontal treatment
- smoking periodontitis (SP): participants who reported smoking >10 cigarettes per day for >5 years with clinical attachment loss ≥3 mm in >30% of sites, with probing depth ≥5 mm in at least six teeth, and with radiographic bone loss extending to or beyond the middle third of the root in the coronal third will be included.
  Interventions: Diagnostic Test: Before non-surgical periodontal treatment; Procedure: non-surgical periodontal treatment; Diagnostic Test: 3rd month after non-surgical periodontal treatment
- non-smoking periodontal health (HC): participants who reported never smoking and periodontal healthy.
  Interventions: Diagnostic Test: Before non-surgical periodontal treatment
- smoking periodontal health (HCS): participants who reported smoking >10 cigarettes per day and periodontal healthy.
  Interventions: Diagnostic Test: Before non-surgical periodontal treatment

INTERVENTIONS:
Diagnostic Test: Before non-surgical periodontal treatment — Clinical Measurements and Laboratory Measurement Saliva and serum samples will be collected from all patients initially. Clinical parameters will also be recorded initially. Plaque index (PI) and gingival index (GI) will be recorded at four sites per tooth. Full-mouth probing depth (PD) and clinical attachment level (CAL) will be detailed per tooth at six sites, and the percentage of bleeding areas will be recorded as present or absent within 20 seconds after probing using a binary scoring system. A calibrated periodontologist (ZTE) will record all clinical parameters using manual probing.
  Following sampling, both serum and saliva samples will be stored at -80°C until analysis. Concentrations of NLRP3, ASC, caspase-1, IL-18, IL-1beta, TNF-alfa, IL-10, TGF-beta, and SIRT-1 will be analyzed by specific enzyme-linked immunosorbent assay (ELISA) kits in both serum and saliva samples. LncRNA SNHG5 and MEG3 will be examined using Real-time PCR.
Procedure: non-surgical periodontal treatment — Treatment will be performed using ultrasonic devices followed by root planing with gracey curettes. SRP will be completed in two visits, each consisting of quadrants every 2 days. Oral hygiene instructions will include demonstrating proper brushing techniques and the use of interdental cleaning aids as needed. Saliva and serum samples will be collected again at the 3-month follow-up visit, all clinical parameter records will be repeated by the same clinician (ZTE), and oral hygiene instructions will be reconfirmed as needed. After the collection of 3-month records and samples, all patients with persistent pockets will be subjected to a standard periodontitis treatment protocol.
  Groups: Non-smoking periodontitis (NSP); smoking periodontitis (SP)
Diagnostic Test: 3rd month after non-surgical periodontal treatment — All clinical and laboratory evaluations described under the heading "Before non-surgical periodontal treatment" will be repeated in the 3rd month after NSPT.
  Groups: Non-smoking periodontitis (NSP); smoking periodontitis (SP)

SUMMARY:
The goal of this observational is to analyze the relationship between levels of interleukin-18 (IL-18), interleukin (IL-1β), Tumor Necrosis Factor-alpha (TNF-α), interleukin-10 (IL-10), transforming growth factor beta (TGF-β), Nucleotide-binding oligomerization domain -like receptor protein 3 (NLRP3), apoptosis-associated speck-like protein (ASC), caspase-1, Sirtuin 1 (SIRT-1), Long noncoding RNA (lncRNA) small nucleolar RNA host gene 5 (SNHG5), and maternally expressed gene 3 (MEG3) in saliva, serum, and peripheral mononuclear blood cell (PMBC)in patients with periodontitis and smokers, to examine the changes in these biomarkers after non surgical periodontal treatment (NSPT), and to evaluate potential confounders that may mediate this relationship.

The main questions it aims to answer are:

question 1: Is there a relationship between the biomarkers mentioned above and periodontitis and smoking? question 2:How do the above-mentioned biomarkers change after NSPT in smokers and non-smokers?

DETAILED DESCRIPTION:
There will be 4 groups in the study: Non-smoking periodontitis (NSP), smoking periodontitis (SP), non-smoking healthy control (HC), and smoking healthy control (HCS).

The periodontitis groups in the study (NSP and SP) will include patients diagnosed with Stage II and III, generalized, Grade B, C periodontitis clinically based on the consensus report of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions, and systemically healthy individuals. Patients with clinical attachment loss ≥3 mm in >30% of sites, with probing depth ≥5 mm in at least six teeth, and with radiographic bone loss extending to or beyond the middle third of the root in the coronal third will be included. Patients with periodontal disease-related tooth loss ≤4 teeth will be included. Disease progression rate will be graded as B or C Class based on direct evidence of disease progression confirmed by panoramic radiographs and evidence of indirect destruction proportional to biofilm accumulations. In the smoking periodontitis group (SP) and smoking healthy group (HCS), participants who reported smoking >10 cigarettes per day for >5 years will be included, while participants in the non-smoking groups (NSP and HC) will be those who reported never smoking.

Clinical Measurements and Non-surgical Periodontal Treatment

Saliva and serum samples will be collected from all patients initially and 3 months after NSPT. Clinical parameters will also be recorded initially and at the 3rd month. Plaque index (PI) and gingival index (GI) will be recorded at four sites per tooth. Full-mouth probing depth (PD) and clinical attachment level (CAL) will be detailed per tooth at six sites, and the percentage of bleeding areas will be recorded as present or absent within 20 seconds after probing using a binary scoring system. A calibrated periodontologist (ZTE) will record all clinical parameters using manual probing. Examiner calibration will be provided before starting the study on a small pilot population to achieve consistent intra-examiner accuracy. After the collection of baseline samples and clinical parameter records, all patients will receive initial periodontal treatment, including patient education, full-mouth scaling, and root planing (SRP), and oral hygiene instructions from the same experienced clinician (ZTE).

Laboratory Measurement

Each patient will be instructed to abstain from eating, drinking, and oral hygiene practices for 12 hours before sampling. Serum and saliva samples will be collected from each patient between 8:00 and 10:00 in the morning before dental examination.

Blood Sampling: In the scope of the study, a total of 5 mL of blood will be collected from the antecubital vein of each individual by an expert nurse from the Department of Periodontology.

For serum sampling, venous puncture will be performed, and blood samples will be collected, immediately cooled on ice, and centrifuged at 4°C (800 rpm for 10 minutes). After the collection of saliva samples, they will be centrifuged immediately at 4°C (1000 rpm for 2 minutes). Following sampling, both serum and saliva samples will be stored at -80°C until analysis. Concentrations of NLRP3, ASC, caspase-1, IL-18, IL-1beta, TNF-alfa, IL-10, TGF-beta, and SIRT-1 will be analyzed by specific enzyme-linked immunosorbent assay (ELISA) kits in both serum and saliva samples. LncRNA SNHG5 and MEG3 will be examined using Real-time polymerase chain reaction (RT-PCR).

IL-18, IL-1beta, TNF-alfa, IL-10, TGF-beta, NLRP3, SIRT-1, lncRNA SNHG5, and MEG3 levels in PMBC will be evaluated using RT-PCR. All analysis steps for each kit will be evaluated using the protocol recommended by the manufacturer.

Statistical Analysis:

Statistical analysis will be performed using commercially available software (SPSS version 22.0, SPSS). In this study, a significance value (p-value) of <0.05 will be used. This study is designed as a prospective controlled clinical trial. The sample size of the study was calculated using the R Statistical Language program (version 4.1.2; The R Foundation for Statistical Computing, Vienna, Austria; http://www.r-project.org). It was planned to include at least 25 individuals in each group for One-Way Analysis of Variance analysis to be conducted with a significance level of 5%, statistical power of 80%, and effect size of 0.4 (Cohen's f=0.4) to determine if there is a significant difference in inflammatory factors between the study groups (smoking periodontitis, smoking periodontally healthy, non-smoking periodontitis, non-smoking periodontally healthy).

Longitudinal analyses will include data only from patients who complete the entire study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65
* Being diagnosed as "periodontally healthy" or "periodontitis" based on periodontal examination
* Not having any accompanying systemic diseases (such as diabetes, cardiovascular diseases, etc.)
* Agreeing to participate in the study

Exclusion Criteria:

* Use of contraceptive medications
* Use of anti-inflammatory, antibiotic, immunosuppressive, or other medications - that could affect the study outcomes within the previous 6 months
* History of excessive alcohol consumption
* Pregnancy or breastfeeding
* Undergoing periodontal treatment within the previous 6 months
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is planned to be conducted with 100 individuals aged between 18 and 65 who apply to the Department of Periodontology, Faculty of Dentistry, Necmettin Erbakan University, for various reasons. The eligibility of individuals to be included in the study will be evaluated by Dr. Zeynep TAŞTAN EROĞLU at the Periodontology Clinic of NEU Faculty of Dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Pre-treatment clinical and laboratory evaluation | baseline
  Comparison of clinical measurements and IL-18, IL-1beta, TNF-alpha, IL-10, TGF-beta, NLRP3, SIRT-1, lncRNA SNHG5, and MEG3 levels of the 4 groups in the study
Comparison of clinical measurements and laboratory measurements at 3 months post-treatment | 3rd month after NSPT
  Comparison of clinical measurements and IL-18, IL-1beta, TNF-alpha, IL-10, TGF-beta, NLRP3, SIRT-1, lncRNA SNHG5, and MEG3 levels of periodontitis groups (NSP and SP) at the 3rd month after treatment